CLINICAL TRIAL: NCT03449147
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, 12-Month Study to Evaluate the Efficacy and Safety of MK-7264 in Adult Participants With Chronic Cough (PN030)
Brief Title: A Study of Gefapixant (MK-7264) in Adult Participants With Chronic Cough (MK-7264-030)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7264-030; MK-7264-030 (Other: Merck Protocol Number); 2017-003559-49 (EudraCT Number)
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Results first posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Chronic Cough
MeSH Terms: conditions — Chronic Cough | interventions — Gefapixant; BID protein, human

STUDY DESIGN:
Intervention Model Description: Participants with refractory or unexplained chronic cough will be randomized to 1 of 3 treatment groups: gefapixant 45 mg twice daily (BID), gefapixant 15 mg BID, or placebo.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive a matching placebo tablet BID during the 24-week main study period and the 28-week extension period.
  Interventions: Drug: Placebo
- Gefapixant 15 mg BID (Experimental): Participants will receive a gefapixant 15 mg tablet BID and placebo tablet to match gefapixant 45 mg BID during the 24-week main study period and the 28-week extension period.
  Interventions: Drug: Placebo; Drug: Gefapixant 15 mg BID
- Gefapixant 45 mg BID (Experimental): Participants will receive a gefapixant 45 mg tablet BID and placebo tablet to match gefapixant 15 mg BID during the 24-week main study period and during the 28-week extension period.
  Interventions: Drug: Placebo; Drug: Gefapixant 45 mg BID

INTERVENTIONS:
Drug: Placebo — Placebo tablet administered orally BID
Drug: Gefapixant 15 mg BID — Gefapixant 15 mg tablet administered orally BID
  Other Names: MK-7264
  Arms: Gefapixant 15 mg BID
Drug: Gefapixant 45 mg BID — Gefapixant 45 mg tablet administered orally BID
  Other Names: MK-7264
  Arms: Gefapixant 45 mg BID

SUMMARY:
The primary objectives of this study are to evaluate the efficacy of gefapixant (MK-7264) in reducing cough frequency as measured over a 24-hour period, and to determine the safety and tolerability of gefapixant. The primary hypothesis is that at least one dose of gefapixant is superior to placebo in reducing coughs per hour (over 24 hours) at Week 24.

DETAILED DESCRIPTION:
This study will have a main 24-week treatment period and a 28-week extension period of treatment (total treatment period of 52 weeks). Participants at selected sites and countries who complete the main and extension study periods may consent to participate in an observational, 12-week, Off-treatment Durability Study Period. Any assessments conducted in the observational period will be exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Chest radiograph or computed tomography scan of the thorax (within 5 years of Screening/Visit 1 and after the onset of chronic cough) not demonstrating any abnormality considered to be significantly contributing to the chronic cough or any other clinically significant lung disease in the opinion of the principal investigator or the sub-investigator
* Has had chronic cough for at least 1 year with a diagnosis of refractory chronic cough or unexplained chronic cough
* Is a female who is not pregnant, not breastfeeding, not of childbearing potential, or agrees to follow contraceptive guidance
* Provides written informed consent and is willing and able to comply with the study protocol (including use of the digital cough recording device and completion of study questionnaires)

Exclusion Criteria:

* Is a current smoker or has given up smoking within 12 months of Screening, or is a former smoker with greater than 20 pack-years
* Has a history of respiratory tract infection or recent clinically significant change in pulmonary status
* Has a history of chronic bronchitis
* Is currently taking an angiotensin converting enzyme inhibitor (ACEI), or has used an ACEI within 3 months of Screening
* Has an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m^2 at Screening OR an eGFR ≥30 mL/min/1.73 m^2 and <50 mL/min/1.73 m^2 at Screening with unstable renal function
* Has a history of malignancy ≤5 years
* Is a user of recreational or illicit drugs or has had a recent history of drug or alcohol abuse or dependence
* Has a history of anaphylaxis or cutaneous adverse drug reaction (with or without systemic symptoms) to sulfonamide antibiotics or other sulfonamide-containing drugs
* Has a known allergy/sensitivity or contraindication to gefapixant
* Has donated or lost ≥1 unit of blood within 8 weeks prior to the first dose of gefapixant
* Has previously received gefapixant
* Currently participating in or has participated in an interventional clinical study within 30 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1317 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (171):
- United States (34):
  - Phoenix Medical Group ( Site 0022), Peoria, Arizona
  - Pulmonary Associates, PA ( Site 0063), Phoenix, Arizona
  - Clinical Research Consortium ( Site 0088), Tempe, Arizona
  - Allergy & Asthma Associates of SCV Research Center ( Site 0064), San Jose, California
  - Lenus Research & Medical Group Llc ( Site 0075), Sweetwater, Florida
  - Atlanta Allergy & Asthma Clinic PA ( Site 0029), Stockbridge, Georgia
  - Rush University Medical Center ( Site 0103), Chicago, Illinois
  - Healthcare Research Network LLC ( Site 0093), Flossmoor, Illinois
  - Abraham Research, PLLC ( Site 0107), Fort Mitchell, Kentucky
  - Paul A. Shapero, MD ( Site 0104), Bangor, Maine
  - Bethesda Allergy Asthma and Research Center LLC ( Site 0019), Bethesda, Maryland
  - Respiratory Medicine Research Institute of Michigan, PLC ( Site 0034), Ypsilanti, Michigan
  - Minnesota Lung Center ( Site 0108), Edina, Minnesota
  - Mayo Clinic - Rochester ( Site 0006), Rochester, Minnesota
  - Minnesota Lung Center ( Site 0041), Woodbury, Minnesota
  - The Lung Research Center ( Site 0072), Chesterfield, Missouri
  - University of Missouri ENT & Allergy Center ( Site 0066), Columbia, Missouri
  - CHI Health Creighton University Medical Center ( Site 0024), Omaha, Nebraska
  - Clinical Research Consortium ( Site 0050), Las Vegas, Nevada
  - Atlantic Research Center LLC ( Site 0012), Ocean City, New Jersey
  - Albuquerque Clinical Trials ( Site 0039), Albuquerque, New Mexico
  - Montefiore Medical Center ( Site 0098), The Bronx, New York
  - Wake Research Associates, LLC ( Site 0058), Raleigh, North Carolina
  - Remington-Davis, Inc. ( Site 0082), Columbus, Ohio
  - Clinical Research Institute of Southern Oregon, PC ( Site 0099), Medford, Oregon
  - Allergy Associates Research Center ( Site 0026), Portland, Oregon
  - AAPRI Clinical Research Institute ( Site 0001), Warwick, Rhode Island
  - Lowcountry Lung & Critical Care, PA ( Site 0045), Charleston, South Carolina
  - Allergic Disease and Asthma Center ( Site 0043), Greenville, South Carolina
  - Clinical Research of Rock Hill ( Site 0079), Rock Hill, South Carolina
  - Clinical Research Partners, LLC. ( Site 0080), Richmond, Virginia
  - Bellingham Asthma & Allergy ( Site 0076), Bellingham, Washington
  - Marycliff Clinical Research ( Site 0062), Spokane, Washington
  - Multicare Health System ( Site 0018), Tacoma, Washington
- Australia (4):
  - Australian Clinical Research Network ( Site 0201), Maroubra, New South Wales
  - Holdsworth House Medical Practice ( Site 0206), Sydney, New South Wales
  - Royal Adelaide Hospital [Adelaide, Australia] ( Site 0214), Adelaide, South Australia
  - Trialswest ( Site 0208), Murdoch
- Canada (8):
  - Hamilton Medical Research Group ( Site 0510), Hamilton, Ontario
  - Recherche GCP Research ( Site 0500), Montreal, Quebec
  - Diex Recherche Quebec Inc ( Site 0515), Québec, Quebec
  - Clinique Specialisee en Allergie de la Capitale - CSAC ( Site 0504), Québec, Quebec
  - Clinique de Pneumologie et du Sommeil de Lanaudiere- CPSL ( Site 0516), Saint-Charles-Borromée, Quebec
  - Q & T Research Sherbrooke Inc. ( Site 0512), Sherbrooke, Quebec
  - CIC Mauricie Inc. ( Site 0503), Trois-Rivières, Quebec
  - Diex Recherche Victoriaville Inc. ( Site 0514), Victoriaville, Quebec
- China (8):
  - The First Affiliated Hospital of Fujian Medical University ( Site 5017), Fuzhou, Fujian
  - The First Affiliated Hospital of Guangzhou Medical University ( Site 5000), Guangzhou, Guangdong
  - Inner Mongolia Autonomous Region Hospital ( Site 5018), Hohhot, Inner Mongolia
  - The First Affiliated Hospital of Nanchang University ( Site 5012), Nanchang, Jiangxi
  - ShengJing Hospital of China Medical University ( Site 5024), Shenyang, Liaoning
  - Shanghai General Hospital ( Site 5010), Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Zhejiang University ( Site 5014), Hangzhou, Zhejiang
  - Peking University Third Hospital ( Site 5005), Beijing
- Colombia (10):
  - Fundacion Centro de Investigacion Clinica CIC ( Site 0603), Medellín, Antioquia
  - Hospital Pablo Tobon Uribe ( Site 0600), Medellín, Antioquia
  - Universidad Pontificia Bolivariana - Clinica Universitaria Bolivariana ( Site 0602), Medellín, Antioquia
  - Neumo Investigaciones SAS ( Site 0622), Bogota, Cundinamarca
  - Centro Especializado en Enfermedades Pulmonares. ( Site 0620), Bogota, Cundinamarca
  - Fundacion Valle del Lili ( Site 0618), Cali, Valle del Cauca Department
  - Centro Medico Imbanaco de Cali S.A ( Site 0619), Cali, Valle del Cauca Department
  - MedPlus Medicina Prepagada S.A. ( Site 0612), Bogotá
  - Instituto Neumologico del Oriente S.A. ( Site 0649), Bucaramanga
  - Inst. Prestadora de Servicios de Salud Universidad Antioquia ( Site 0621), Medellín
- Czechia (5):
  - MUDr. I. Cierna Peterova s.r.o. ( Site 0707), Brandýs nad Labem
  - MediTrial s.r.o ( Site 0702), Jindrichuv Hradec III
  - Ordinace Pneumologie a diagnostiky Plicnich funkci ( Site 0705), Karlovy Vary
  - PNEUMO-NB s.r.o. ( Site 0710), Nový Bor
  - Nemocnice Tabor a.s. ( Site 0703), Tábor
- Denmark (2):
  - Herlev Hospital ( Site 0803), Herlev
  - Bispebjerg Hospital ( Site 0804), København NV
- Germany (7):
  - Aerztezentrum Axel Springer Passage ( Site 1009), Berlin
  - Atemwegszentrum Neukoeln ( Site 1003), Berlin
  - Gemeinschaftspraxis Zentrum ( Site 1005), Frankfurt
  - Pneumologicum im Suedstadtforum ( Site 1004), Hanover
  - Pneumologenzentrum ( Site 1006), Leipzig
  - Ballenberger Freytag Wenisch Institut fuer klinische Forschung GmbH ( Site 1011), Neu-Isenburg
  - PneumoConsult Ulm ( Site 1008), Ulm
- Guatemala (5):
  - Clinipharm ( Site 2902), Guatemala City
  - Celan SA ( Site 2900), Guatemala City
  - Consultorio Privado Dr. Jeremias Guerra ( Site 2909), Guatemala City
  - Clinica Medica Especializada en Neumologia ( Site 2901), Guatemala City
  - Clinica Privada Dr. Jose Francisco Flores Lopez ( Site 2903), Guatemala City
- Hungary (8):
  - Dr Kenessey Albert Korhaz-Rendelointezet ( Site 1200), Balassagyarmat
  - Synexus Magyarorszag Kft. ( Site 1208), Budapest
  - Erzsebet Gondozohaz ( Site 1207), Gödöllő
  - Synexus Magyarorszag Kft. ( Site 1210), Gyula
  - Lumniczer Sandor Korhaz es Rendelointezet ( Site 1212), Kapuvár
  - CRU Hungary KFT ( Site 1205), Miskolc
  - Da Vinci Private Clinic - Da Vinci Maganklinika ( Site 1201), Pécs
  - Puspokladanyi Egeszsegugyi Szolgaltato Nonprofit Kft ( Site 1203), Püspökladány
- Kaplan Medical Center ( Site 1300), Rehovot, Israel
- Azienda Ospedaliero Universitaria Careggi ( Site 1400), Florence, Italy
- Malaysia (6):
  - Hospital Sultanah Bahiyah ( Site 1607), Alor Star, Kedah
  - Hospital Taiping ( Site 1600), Taiping, Perak
  - Hospital Pulau Pinang. ( Site 1606), George Town, Pulau Pinang
  - Universiti Teknologi MARA ( Site 1602), Batu Caves, Selangor
  - Institut Perubatan Respiratori ( Site 1605), Kuala Lumpur
  - University Malaya Medical Centre ( Site 1601), Kuala Lumpur
- New Zealand (4):
  - Southern Clinical Trials - Waitemata ( Site 0230), Auckland
  - Middlemore Clinical Trials ( Site 0232), Auckland
  - Lakeland Clinical Trials ( Site 0233), Rotorua
  - P3 Research Ltd. ( Site 0228), Tauranga
- Peru (5):
  - Clinica Ricardo Palma ( Site 1802), San Isidro, Lima region
  - Hospital Nacional Adolfo Guevara Velasco ( Site 1808), Cusco
  - Clinica Internacional ( Site 1801), Lima
  - Asociacion Civil por la Salud ( Site 1805), Lima
  - Hospital Nacional Cayetano Heredia [Lima, Peru] ( Site 1806), Lima
- Poland (14):
  - NZOZ CENTRUM ALERGOLOGII ( Site 1909), Lublin, Lublin Voivodeship
  - Centrum Medyczne Pratia Katowice ( Site 1917), Katowice, Silesian Voivodeship
  - Centrum Medyczne Silmedic Sp z o o ( Site 1920), Katowice, Silesian Voivodeship
  - Centrum Medycyny Oddechowej Mroz Spolka Jawna ( Site 1918), Bialystok
  - KLIMED ( Site 1902), Bychawa
  - Gyncentrum Clinic Sp. z o.o. ( Site 1908), Katowice
  - Specjalistyczny osrodek .All-Med. Grazyna Pulka ( Site 1919), Krakow
  - Centrum Nowoczesnych Terapii Dobry Lekarz ( Site 1924), Krakow
  - Uniwersytecki Szpital Kliniczny im. Norberta Barlickiego nr 1 ( Site 1921), Lodz
  - Ostrowieckie Centrum Medyczne ( Site 1915), Ostrowiec Świętokrzyski
  - RCMed ( Site 1912), Sochaczew
  - Lubelskie Centrum Diagnostyczne ( Site 1913), Świdnik
  - Centrum Medyczne Pratia Warszawa ( Site 1911), Warsaw
  - Centrum Medyczne Lucyna Andrzej Dymek - Zawadzkie ( Site 1923), Zawadzkie
- South Africa (7):
  - Iatros International ( Site 2130), Brandwag, Bloemfontein
  - Rochester Place Medical Centre ( Site 2129), Morningside, Gauteng
  - Jongaie Research ( Site 2131), Pretoria, Gauteng
  - Dr N K Gounden Mediclinic ( Site 2134), Shallcross, KwaZulu-Natal
  - Drs Lalloo & Ambaram ( Site 2132), Umhlanga Ridge, KwaZulu-Natal
  - I Engelbrecht Research ( Site 2128), Centurion, Tswane
  - UCT Lung Institute - Bateman ( Site 2126), Cape Town, Western Cape
- Turkey (Türkiye) (9):
  - Uludag Universitesi Tip Fakultesi ( Site 2621), Bursa, Gorukle
  - Cukurova Universitesi Tıp Fakultesi Balcalı Hastanesi ( Site 2612), Adana
  - Ankara Universitesi Tip Fakultesi Cebeci Hastanesi ( Site 2602), Ankara
  - Trakya Universitesi Saglik Arastirma ve Uygulama Merkezi ( Site 2619), Edirne
  - Istanbul Universitesi Istanbul Tip Fakultesi Gogus Hastalıklari ABD ( Site 2610), Istanbul
  - SSK Sureyyapasa Gogus Hastaliklari Hastanesi ( Site 2608), Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi ( Site 2603), Izmir
  - SBU Dr. Suat Seren Gogus Hast. ve Cer. Egitim ve Arastirma Hast. ( Site 2604), Izmir
  - Celal Bayar University Faculty of Medicine ( Site 2614), Manisa
- Ukraine (15):
  - Chernihiv City hospital N2 ( Site 2801), Chernihiv
  - CE Chernivtsi state city clinical hospital 3 ( Site 2806), Chernivtsi
  - Kherson City Clinical Hospital n.a. Y.Y. Karabelesh ( Site 2812), Kherson
  - Medical Clinic Blagomed LLC ( Site 2807), Kiev
  - Kyiv City Tuberculosis Hospital No. 1 ( Site 2814), Kyiv
  - Medical Association Medbud of the PJSC Kyivmiskbud ( Site 2803), Kyiv
  - SE Road Clinical Hospital 2 of Kyiv station ( Site 2809), Kyiv
  - Institute of Otolaryngology n. a. Prof. A. I. Kolomiychenko ( Site 2833), Kyiv
  - F.G.Yanovskyy Institute of Phthisiology and Pulmonology ( Site 2804), Kyiv
  - F.G.Yanovskyy Institute of Phthisiology and Pulmonology ( Site 2830), Kyiv
  - Volyn Regional Clinical Hospital ( Site 2829), Lutsk
  - Poltava City Clinical Hospital 1 ( Site 2808), Poltava
  - Vinnytsia Regional Clinical Hospital n.a. M.I. Pyrogov ( Site 2819), Vinnytsia
  - MI Zaporizhzhia City Multispecialty Clinical Hospital 9 ( Site 2811), Zaporizhzhia
  - Zhytomyr Central City Hospital #1 ( Site 2828), Zhytomyr
- United Kingdom (18):
  - Hull & East Yorkshire NHS Trust. Castle Hill Hospital ( Site 2704), Cottingham, East Yorkshire
  - Synexus Midlands Clinical Research Centre Ltd ( Site 2719), Birmingham, Edgbaston
  - Medinova East London Dedicated Research Centre ( Site 2715), Romford, Essex
  - Medinova South London Dedicated Research Centre ( Site 2714), Sidcup, Kent
  - Medinova North London Dedicated Research Centre ( Site 2716), Northwood, Middlesex
  - Medinova Lakeside Dedicated Research Centre ( Site 2710), Corby, Northamptonshire
  - Medinova Warwickshire Dedicated Research Centre ( Site 2717), Kenilworth, Warwickshire
  - Belfast City Hospital ( Site 2705), Belfast
  - Synexus Scotland Clinical Research Centre ( Site 2721), Glasgow
  - Synexus Merseyside Clinical Research Centre ( Site 2720), Liverpool
  - Prince Phillip Hospital ( Site 2722), Llanelli
  - 1Kings College Hospital ( Site 2702), London
  - Synexus Manchester Clinical Research Centre ( Site 2718), Manchester
  - Wythenshawe Hospital ( Site 2700), Manchester
  - North Tyneside General Hospital ( Site 2707), North Shields
  - Rothwell Medical Centre ( Site 2712), Rothwell
  - Taunton and Somerset Hospital ( Site 2723), Taunton
  - West Walk Surgery ( Site 2711), Yate

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Dicpinigaitis PV, Birring SS, Blaiss M, McGarvey LP, Morice AH, Pavord ID, Satia I, Smith JA, La Rosa C, Li Q, Nguyen AM, Schelfhout J, Tzontcheva A, Muccino D. Demographic, clinical, and patient-reported outcome data from 2 global, phase 3 trials of chronic cough. Ann Allergy Asthma Immunol. 2023 Jan;130(1):60-66. doi: 10.1016/j.anai.2022.05.003. Epub 2022 May 13. PMID 35569802
- [Derived] McGarvey LP, Birring SS, Morice AH, Dicpinigaitis PV, Pavord ID, Schelfhout J, Nguyen AM, Li Q, Tzontcheva A, Iskold B, Green SA, Rosa C, Muccino DR, Smith JA; COUGH-1 and COUGH-2 Investigators. Efficacy and safety of gefapixant, a P2X3 receptor antagonist, in refractory chronic cough and unexplained chronic cough (COUGH-1 and COUGH-2): results from two double-blind, randomised, parallel-group, placebo-controlled, phase 3 trials. Lancet. 2022 Mar 5;399(10328):909-923. doi: 10.1016/S0140-6736(21)02348-5. PMID 35248186

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1317 participants were randomized to the 52-week treatment period, and 1314 participants received at least 1 dose of study intervention. After the main study, 122 participants continued in an optional Off-Treatment observational study period (no treatment).
Groups:
- Placebo: Participants received dose-matched placebo tablets twice daily (BID) during the 24-week main study period and 28-week extension period.
- Gefapixant 15 mg BID: Participants received a gefapixant 15 mg tablet and placebo tablet to match gefapixant 45 mg BID during the 24-week main study period and 28-week extension period.
- Gefapixant 45 mg BID: Participants received a gefapixant 45 mg tablet and placebo tablet to match gefapixant 15 mg BID during the 24-week main study period and 28-week extension period.
Period: 52-week Treatment Period
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Started | 436 | 442 | 439
Completed | 382 | 368 | 355
Not Completed | 54 | 74 | 84
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 6 | 2 | 5
Not completed — Other | 0 | 1 | 2
Not completed — Physician Decision | 1 | 0 | 3
Not completed — Screen Failure | 1 | 2 | 0
Not completed — Withdrawal by Subject | 46 | 68 | 74
Period: 12-Week Off-Treatment Durability Period
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Started | 48 (Not all participants continued in the optional Off-Treatment Period.) | 37 (Not all participants continued in the optional Off-Treatment Period.) | 37 (Not all participants continued in the optional Off-Treatment Period.)
Completed | 47 | 36 | 37
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID | Total
Number analyzed (Participants) | 436 | 442 | 439 | 1317
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (12.5) | 58.4 (11.3) | 57.8 (12.4) | 58.2 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 326 | 331 | 329 | 986
  Male | 110 | 111 | 110 | 331
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 85 | 93 | 89 | 267
  Not Hispanic or Latino | 348 | 347 | 344 | 1039
  Unknown or Not Reported | 3 | 2 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 20 | 28 | 24 | 72
  Asian | 15 | 14 | 15 | 44
  Native Hawaiian or Other Pacific Islander | 4 | 2 | 3 | 9
  Black or African American | 5 | 9 | 14 | 28
  White | 356 | 358 | 346 | 1060
  More than one race | 36 | 31 | 37 | 104
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline 24-Hour Coughs Per Hour [Mean (Standard Deviation); unit: Coughs/Hour] — 24-hour coughs per hour is defined as the average hourly cough frequency based on 24-hour sound recordings using a digital recording device (cough monitor). Population: All participants with 24-hour coughs per hour data available at baseline
  Coughs/Hour
    number analyzed (Participants) | 432 | 431 | 434 | 1297
    (all) | 27.45 (24.44) | 26.82 (21.25) | 26.84 (27.04) | 27.04 (24.35)

OUTCOME MEASURES:

1. Primary Outcome: Model-Based Geometric Mean Ratio (GMR) of 24-Hour Coughs Per Hour at Week 24/Baseline
Description: 24-hour coughs per hour was defined as the average hourly cough frequency based on 24-hour sound recordings using a digital recording device (cough monitor). A longitudinal analysis of covariance (ANCOVA) model was applied to log-transformed cough data to determine geometric mean (GM) 24-hour coughs per hour at baseline and week 24. The GMR (Week 24 GM 24-hour coughs per hour divided by Baseline GM 24-hour coughs per hour) is reported.
Time Frame: Baseline, Week 24
Population: All randomized participants who took at least 1 dose of study intervention, had available 24-hour cough data at baseline and at least one available post-baseline measurement during the treatment period.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Number analyzed (Participants) | 419 | 415 | 409
Ratio | 0.43 [0.39 to 0.48] | 0.43 [0.38 to 0.47] | 0.37 [0.33 to 0.41]
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 15 mg BID; Estimated relative reduction (ERR) relative to Placebo (i.e. estimated percent change difference) was calculated by 100 (e**DIFF -1), where e = exponent of difference; and DIFF= treatment difference in change from baseline at Week 24 based on log transformed data; Test type: Superiority; p = 0.875, ANCOVA — Comparison based on a longitudinal ANCOVA model that included treatment, visit, treatment-by-visit interaction, gender, region, log-transformed baseline value, and log-transformed baseline value-by-visit as covariates; Estimated Relative Reduction (%) = -1.14, 95% CI 2-sided [-14.27 to 14.02]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 45 mg BID; ERR relative to Placebo (i.e. estimated percent change difference) was calculated by 100 (e**DIFF -1), where e = exponent of difference; and DIFF= treatment difference in change from baseline at Week 24 based on log transformed data; Test type: Superiority; p = 0.031, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Estimated Relative Reduction (%) = -14.64, 95% CI 2-sided [-26.07 to -1.43]

2. Primary Outcome: Number of Participants Who Experienced At Least One Adverse Event (AE) During Treatment and Follow-up
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Time Frame: Up to 54 Weeks
Population: All randomized participants who received at least one dose of study intervention during the 52-week treatment period. Per protocol, participants in the optional off-treatment observational period were not included. 3 participants randomized to placebo group who took 1 or more incorrect dose(s) of study drug were counted in the higher dose group of gefapixant received: 2 participants were analyzed in the gefapixant 15 mg group and 1 was analyzed in the gefapixant 45 mg group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Number analyzed (Participants) | 432 | 442 | 440
Participants | 349 | 373 | 399

3. Primary Outcome: Number of Participants Who Discontinued a Study Drug Due to an AE
Description: as for outcome 2
Time Frame: Up to 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Number analyzed (Participants) | 432 | 442 | 440
Participants | 25 | 40 | 100

4. Secondary Outcome: Model-Based GMR of Awake Coughs Per Hour at Week 24/Baseline
Description: Awake coughs per hour was defined as the average hourly cough frequency while the participant is awake, based on a 24-hour interval of sound recordings using a digital recording device (cough monitor). ANCOVA model was applied to log-transformed cough data to determine GM of awake coughs per hour at baseline and week 24. The GMR (Week 24 GM awake coughs per hour divided by Baseline GM awake coughs per hour) is reported.
Time Frame: Baseline, Week 24
Population: All randomized participants who took at least 1 dose of study intervention, had available awake 24-hour cough data at baseline and at least one available post-baseline measurement during the treatment period.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Number analyzed (Participants) | 419 | 415 | 409
Ratio | 0.42 [0.38 to 0.47] | 0.41 [0.37 to 0.46] | 0.36 [0.32 to 0.40]
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 15 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.677, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Estimated Relative Reduction (%) = -3.03, 95% CI 2-sided [-16.14 to 12.12]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 45 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.022, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Estimated Relative Reduction (%) = -15.79, 95% CI 2-sided [-27.27 to -2.50]

5. Secondary Outcome: Percentage of Participants With a ≥1.3 Point Change From Baseline in the Leicester Questionnaire (LCQ) Total Score at Week 24
Description: The 19-item LCQ assessed the impact of chronic cough in three health-related quality of life (HRQoL) domains (physical, social and psychological). The LCQ is calculated as a mean score for each domain ranging from 1 to 7, with a total score ranging from 3 to 21. Higher scores indicate better HRQoL. A clinically meaningful improvement from baseline in HRQoL was defined as ≥1.3-point increase in the LCQ total score at Week 24. The percentage of participants (logistic regression model-based) with a ≥1.3-point increase in the LCQ total score at Week 24 is presented.
Time Frame: Baseline, Week 24
Population: All randomized participants who had taken at least 1 dose of study intervention, had available LCQ data at baseline, and at least one available post-baseline measurement in the treatment period.
Measure: Number; unit: Percentage of Participants
Groups:
- Gefapixant 45 mg: Participants received a gefapixant 45 mg tablet and placebo tablet to match gefapixant 15 mg BID during the 24-week main study period and 28-week extension period.
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg
Number analyzed (Participants) | 406 | 404 | 399
Percentage of Participants | 70.1 | 75.9 | 76.8
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 15 mg BID; Test type: Superiority; p = 0.077, Regression, Logistic — Comparison based on logistic regression model that included treatment, visit, treatment-by-visit interaction, gender, region, baseline LCQ total score, and the interaction of baseline LCQ total score by visit as covariates; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.97 to 1.85]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 45 mg; Test type: Superiority; p = 0.040, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.02 to 1.96]

6. Secondary Outcome: Percentage of Participants With a ≤-30% Change From Baseline in 24-hour Coughs Per Hour at Week 24
Description: 24-hour coughs per hour was defined as the average hourly cough frequency based on 24-hour sound recordings using a digital recording device (cough monitor). A clinically meaningful improvement from baseline is defined as a ≤-30% change (≥30% reduction) in 24-hour coughs per hour at week 24. The percentage of participants (logistic regression model-based) with a ≤ -30% change from baseline in 24-hour coughs per hour at Week 24 (≥30% reduction from baseline) is presented.
Time Frame: Baseline, Week 24
Population: All randomized participants who took at least 1 dose of study intervention, had available 24-hour cough data at baseline and at least one available post-baseline measurement in the treatment period.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Number analyzed (Participants) | 419 | 415 | 409
Percentage of Participants | 66.9 | 67.4 | 72.9
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 15 mg BID; Test type: Superiority; p = 0.872, Regression, Logistic — Comparison based on a logistic regression model that included treatment, visit, treatment-by-visit interaction, gender, region, baseline 24-hour coughs per hour and the interaction of baseline 24-hour coughs per hour as covariates; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.75 to 1.40]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 45 mg BID; Test type: Superiority; p = 0.082, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.96 to 1.83]

7. Secondary Outcome: Percentage of Participants With ≤-1.3 Point Change From Baseline of Mean Weekly Cough Severity Diary (CSD) Total Score at Week 24
Description: The 7-item CSD was used to record participants' daily cough frequency, cough intensity, and disruption due to cough. Each item was rated on an 11-point scale ranging from 0 (best) to 10 (worst); the total daily CSD score was the sum of these seven item scores (Min=0, Max=70). Mean weekly CSD total score was defined as the average of the mean total daily scores collected during the week prior to each visit. The percentage of participants (logistic regression model-based) with a ≤-1.3 point change from baseline in CSD at Week 24 (or ≥1.3 point reduction from baseline) is reported.
Time Frame: Baseline, Week 24
Population: All randomized participants who had taken at least 1 dose of study intervention, had available CSD data at baseline, and at least one available post-baseline measurement in the treatment period.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg
Number analyzed (Participants) | 428 | 426 | 425
Percentage of Participants | 69.1 | 74.8 | 77.1
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 15 mg BID; Comparison based on a logistic regression model that included treatment, visit, treatment-by-visit interaction, gender, region, baseline mean weekly CSD total score, and the interaction of baseline mean weekly CSD total score by visit as covariates; Test type: Other; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.96 to 1.83]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 45 mg; [analysis description as in outcome 7, analysis 1]; Test type: Other; Odds Ratio (OR) = 1.50, 95% CI 2-sided [1.08 to 2.09]

8. Secondary Outcome: Percentage of Participants With ≤-2.7 Point Change From Baseline of Mean Weekly CSD Total Score at Week 24
Description: The 7-item CSD was used to record participants' daily cough frequency, cough intensity, and disruption due to cough. Each item was rated on an 11-point scale ranging from 0 (best) to 10 (worst); the total daily CSD score was the sum of these seven item scores (Min=0, Max=70). Mean weekly CSD total score was defined as the average of the mean total daily scores collected during the week prior to each visit. The percentage of participants (logistic regression model-based) with a ≤-2.7 point change from baseline in CSD at Week 24 (or ≥2.7 point reduction from baseline) is reported.
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg
Number analyzed (Participants) | 428 | 426 | 425
Percentage of Participants | 41.0 | 46.6 | 55.2
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 15 mg BID; [analysis description as in outcome 7, analysis 1]; Test type: Other; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.93 to 1.69]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 45 mg; [analysis description as in outcome 7, analysis 1]; Test type: Other; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.31 to 2.39]

9. Secondary Outcome: Percentage of Participants With a ≤-30 Millimeter (mm) Change From Baseline in Cough Severity Visual Analog Scale (VAS) Score at Week 24
Description: The VAS is a single-item questionnaire with the response on a 100- point scale ranging from 0 ("No Cough") to 100 ("Extremely Severe Cough"). Mean weekly VAS score was defined as the average of the VAS scores collected during the week prior to each visit. The percentage of participants (logistic regression model-based) with a ≤-30 mm change from baseline in cough severity VAS score at Week 24 is reported.
Time Frame: Baseline, Week 24
Population: All randomized participants who had taken at least 1 dose of study intervention, had available VAS data at baseline, and at least one available post-baseline measurement in the treatment period.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg
Number analyzed (Participants) | 428 | 426 | 425
Percentage of participants | 40.9 | 51.4 | 53.3
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 15 mg BID; Comparison based on a logistic regression model that included treatment, visit, treatment-by-visit interaction, gender, region, baseline mean weekly VAS score, and the interaction of baseline mean weekly VAS score by visit as covariates; Test type: Other; Odds Ratio (OR) = 1.53, 95% CI 2-sided [1.14 to 2.05]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 45 mg; [analysis description as in outcome 9, analysis 1]; Test type: Other; Odds Ratio (OR) = 1.65, 95% CI [1.23 to 2.22]

ADVERSE EVENTS:
Time Frame: On-Treatment Period: Up to Week 54; Off-Treatment (Off-Tx) Period: From Week 52 through Week 64 (approximately 12 weeks)
Description: All-cause mortality (ACM) includes all randomized participants; serious and other AEs include all randomized participants who took ≥1 one dose of study drug. In the treatment period, 3 participants randomized to placebo who took ≥1 incorrect dose(s) of study drug were counted as follows: 2 participants were analyzed in the gefapixant 15 mg arm and 1 in the gefapixant 45 mg arm. AEs and ACM were reported separately for the Treatment Period (MedDRA 23.0) and Off-Tx Period (MedDRA 23.1).
Groups:
- Placebo: Off Tx: Participants previously treated with dose-matched placebo BID for 52 weeks during the main study and extension study periods were observed for up to 3 months during an optional Off-Treatment Durability study period (participants received no treatment).
- Gefapixant 15 mg BID: Off Tx: Participants previously treated with gefapixant 15 mg BID for 52 weeks during the main study and extension study periods were observed for up to 3 months during an optional Off-Treatment Durability study period (participants received no treatment).
- Gefapixant 45 mg BID: Off Tx: Participants previously treated with gefapixant BID for 52 weeks during the main study and extension study periods were observed for up to 3 months during an optional Off-Treatment Durability study period (participants received no treatment).
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID | Placebo: Off Tx | Gefapixant 15 mg BID: Off Tx | Gefapixant 45 mg BID: Off Tx
All-Cause Mortality (participants affected / at risk) | 0/433 | 1/444 | 0/440 | 0/48 | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 25/432 | 24/442 | 25/440 | 0/48 | 0/37 | 1/37
Other Adverse Events (participants affected / at risk) | 248/432 | 290/442 | 359/440 | 6/48 | 3/37 | 1/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=432) | Gefapixant 15 mg BID (N=442) | Gefapixant 45 mg BID (N=440) | Placebo: Off Tx (N=48) | Gefapixant 15 mg BID: Off Tx (N=37) | Gefapixant 45 mg BID: Off Tx (N=37)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital choroid plexus cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disinfectant poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=432) | Gefapixant 15 mg BID (N=442) | Gefapixant 45 mg BID (N=440) | Placebo: Off Tx (N=48) | Gefapixant 15 mg BID: Off Tx (N=37) | Gefapixant 45 mg BID: Off Tx (N=37)
Diarrhoea (Gastrointestinal disorders) | 18 (20) | 27 (29) | 27 (34) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 11 (12) | 15 (15) | 32 (34) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 32 (42) | 26 (33) | 47 (57) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 23 (27) | 20 (24) | 18 (19) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 35 (45) | 29 (35) | 24 (27) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 70 (101) | 93 (128) | 70 (95) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 18 (20) | 23 (25) | 14 (16) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 26 (32) | 38 (47) | 30 (39) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 23 (27) | 34 (40) | 19 (26) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (37) | 22 (26) | 21 (25) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (33) | 30 (34) | 16 (17) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 6 (6) | 13 (14) | 67 (75) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 28 (30) | 56 (64) | 193 (220) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 67 (128) | 74 (131) | 70 (131) | 1 (1) | 0 (0) | 0 (0)
Hypogeusia (Nervous system disorders) | 3 (3) | 17 (18) | 60 (60) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 8 (8) | 37 (39) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 13 (18) | 19 (29) | 1 (1) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 30 (37) | 31 (38) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 13 (13) | 23 (24) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT03449147/Prot_SAP_000.pdf